CLINICAL TRIAL: NCT03688971
Title: A Phase 2, Randomized, Vehicle and Ketoconazole-Controlled, Evaluator-Blinded, Study to Explore the Efficacy, Pharmacodynamics and Safety of Omiganan 1.75% Topical Gel BID in Patients With Mild to Moderate Facial Seborrheic Dermatitis
Brief Title: Omiganan Twice a Day (BID) in Patients With Facial Seborrheic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-017
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — Omiganan; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Omiganan Topical Gel (Experimental): Omiganan 1.75%
  Interventions: Drug: Omiganan
- Ketoconazole Topical Cream (Active Comparator): Ketoconazole 2.0%
  Interventions: Drug: Ketoconazole
- Vehicle (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omiganan — Omiganan Topical Gel
  Arms: Omiganan Topical Gel
Drug: Ketoconazole — Ketoconazole Cream
  Arms: Ketoconazole Topical Cream
Drug: Placebo — Vehicle
  Arms: Vehicle

SUMMARY:
To explore the efficacy and pharmacodynamic effects of omiganan topical gel in facial seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with mild to moderate facial SD (IGA 2 or 3), ≥18 years of age, inclusive. The health status is verified by absence of evidence of any clinical significant active or uncontrolled chronic disease other than SD following a detailed medical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, virology and urinalysis;
* Confirmed SD diagnosis by dermatologist
* Significant facial SD affected area as judged by the investigator or medically qualified designee
* Able to participate and willing to give written informed consent and to comply with the study restrictions;
* Willing to refrain from using other SD treatments in the local treatment area
* Subjects and their partners of childbearing potential must use effective contraception, for the duration of the study and for 3 months after the last dose.

Exclusion Criteria:

* Any current and / or recurrent clinical significant skin condition other than SD;
* Ongoing use of prohibited SD medication. Washout periods prior to baseline are as follows;

  1. Topical steroids, antibiotics, antifungals or other topical (OTC) therapies: 2 weeks
  2. Systemic steroids, antibiotics, antifungals or other systemic therapies: 4 weeks;
  3. Phototherapy: 3 weeks;
  4. Regular use of shampoo for the treatment of PC (including but not limited to OTC zinc pyrithione shampoo), soap for the treatment of seborrheic dermatitis: 2 weeks
  5. Changing a soap, method for daily facial and hair washing: 1 week
* Known hypersensitivity to the compounds or excipients of the compounds;
* Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks of enrollment;
* Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding;
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times in the past year;
* Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Seborrheic dermatitis area severity index (SDASI) | 6 Weeks
  Assessment of erythema, scales and papules and each are scored as 0=none to 3=severe.
Investigator global assessment (IGA) | 6 Weeks
  This is a 5-point scale ranging from 0=clear to 4=severe.
Area of involvement | 6 Weeks
  Facial area involvement is estimated as a % of the body surface area (BSA)
Patient Reported Outcome (PRO) - eDiary | 4 Weeks
  Single-question assessment regarding patient's worst itch. On a scale of 0-100, 0=no itch and 100=worst itch.
PRO - 5-D itch scale | 6 Weeks
  Multidimensional measure of itching. Covers 5 domains: duration, degree, direction, disability and distribution.
PRO - dermatology life quality index (DLQI) | 6 Weeks
  Asses health-related quality of life in general dermatology disability index
Standardized photography | 6 Weeks
  Facial photographs will be taken by a 2D camera (VISIA-CR)
Sebum measurements | 6 Weeks
  Measurement of sebum excretion by Sebumeter
Trans Epidermal Water Loss (TEWL) | 6 Weeks
  To assess barrier status of lesional and non-lesional skin.
Optical Coherence Tomography (OCT) | 6 Weeks
  Measurement of cutaneous morphology of seborrheic dermatitis
Liquid chromatography-mass spectrometry (LC-MS) | 6 Weeks
  Will evaluate the changes in lipid composition of stratum corneum (SC).

SECONDARY OUTCOMES:
Skin microbiota | 6 Weeks
  collection of skin culture sample to evaluate skin microbiota
Skin mycobiota | 6 Weeks
  collection of skin culture sample to evaluate skin mycobiota
Faecal microbiome | 4 Weeks
  collection of faecal samples to evaluate faecal microbiome
Adverse events collected throughout the study | 6 Weeks
Vital signs performed at screening and end of study | 6 Weeks
  Evaluation of systolic and diastolic blood pressure
Vital signs performed at screening and end of study | 6 Weeks
  Evaluation of pulse rate
Vital signs performed at screening and end of study | 6 Weeks
  Evaluation of temperature
12-Lead ECGs performed at screening and end of study | 6 Weeks
  Assessment of heart rate
12-Lead ECGs performed at screening and end of study | 6 Weeks
  Assessment of PR, QRS, QT, QTcB and QTcF
Haematology blood sample assessment | 6 Weeks
  Evaluation of blood collected in BD Vacutainer K2EDTA tube.
Chemistry blood sample assessment | 6 Weeks
  Evaluation of blood collected in BD Vacutainer SST Gel and Clot Activator tube.
Urinalysis urine sample assessment | 6 Weeks
  Evaluation of urine specimen by dipstick
Collection of concomitant medications | 6 Weeks
  questionnaire at each visit to collect concomitant medications taken

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands